CLINICAL TRIAL: NCT02006745
Title: Open Label, Randomised, Pilot Trial of Pegylated Interferon, Ribavirin & Telaprevir vs Pegylated Interferon & Ribavirin Alone in Response Guided Treatment of Acute Hepatitis C Genotype 1 Virus Infection in Patients With HIV-1 Co-infection
Brief Title: Open Label Trial of PEG-IFN, RBV & TVR vs. PEG-IFN & RBV Alone in Tx of HCV-1 in HIV-1 Co-infected Patients (CHAT)
Acronym: CHAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SSAT 052
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: HIV
MeSH Terms: interventions — Ribavirin; telaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ribavirin (Other): ARM 1: PEG-IFN and weight-based ribavirin (RBV)
  Interventions: Drug: Ribavirin
- Telaprevir (Other): ARM 2: PEG-IFN and weight-based RBV plus telaprevir (TPV)
  Interventions: Drug: Telaprevir

INTERVENTIONS:
Drug: Ribavirin — 24 weeks in those achieving RVR (undetectable HCV RNA at 4 weeks) or 48 weeks in those not achieving RVR
  Other Names: PEG-IFN and weight-based ribavirin (RBV)
  Arms: Ribavirin
Drug: Telaprevir — 12 weeks in those achieving RVR, 24 weeks in those not achieving RVR (HCV RNA >25 but <1000 iU/mL at week 4) or 48 weeks in those not achieving RVR (HCV RNA >1000 iU/mL at week 4).
  Other Names: -ARM 2: PEG-IFN and weight-based RBV plus telaprevir (TPV)
  Arms: Telaprevir

SUMMARY:
The purpose of the study is to explore the treatment of patients with acute hepatitis C infection (infection acquired within the last 6 months) who are also infected with human immunodeficiency virus (HIV).

DETAILED DESCRIPTION:
In this study, we will compare two treatment options for hepatitis C in patients who also have HIV infection, to see if there are any differences in the numbers of patients treated who successfully got rid of the hepatitis C virus when the treatment was complete. We will also compare how well the two treatment options are tolerated by the patients taking them.

ELIGIBILITY:
Inclusion Criteria:

* 1. Is male or female aged 18 years or above 2. Has signed the Informed Consent Form voluntarily 3. Documented current acute hepatitis C genotype 1 infection with detectable HCV-RNA (PCR-assay) with an estimated duration less than 24 weeks as defined below:

  1. HCV RNA positive AND
  2. Prior negative anti-HCV antibody or HCV RNA test within 6 months OR
  3. rise of liver transaminases above 2.5 x ULN within the past 6 months with prior normal transaminases during the year before AND
  4. exclusion of other causes of acute hepatitis 4. Confirmed HIV infection 5. Receiving a atazanavir- or efavirenz- or raltegravir-based ART regimen or able to switch regimen to these agents with an undetectable HIV viral load for at least 3 months, or not receiving ART with no immediate plans to start ART during the first 6 months of study 6. CD4 T cell count >200/µl at screening in patients under ART, CD4 T cell count >500/µl at screening in patients without ART 7. If female and of childbearing potential, is using effective birth control methods (as agreed by the investigator) and is willing to continue practising these birth control methods during the trial and for at least 4 months after the last dosage of ribavirin (ie 4 months after week 12, 24 or 48, depending on study arm and treatment response). Routine monthly pregnancy tests must also be performed during this time. Note: Women who are postmenopausal for least 2 years, women with total hysterectomy, and women who have a tubal ligation are considered of non-childbearing potential 8. Heterosexually active male participants or their female partners must use effective birth control methods (as agreed by the investigator) during the trial and for at least 7 months after the last dosage of ribavirin (ie 7 months after week 12, 24 or 48, depending on study arm and treatment response).

Exclusion Criteria:

* . HCV infection with non-1 genotype 2. Acute opportunistic infection requiring treatment 3. Malignancy requiring chemotherapy or radiotherapy 4. Active HBV infection (HBs Ag + with positive hepatitis B DNA) 5. Known autoimmune disease 6. Hepatic failure 7. History of ischaemic heart disease or other serious cardiac disease 8. Serious psychiatric disease which in the view of the investigator precludes the use of interferon 9. Haemoglobinopathy or severe anaemia of any cause 10. Serious abnormality on screening blood tests including, but not limited to: Hemoglobin <10g/dl, absolute neutrophil count <1000/mm3, platelets <90,000/mm3, creatinine clearance <60ml/min 11. If female, she is pregnant or breastfeeding 12. Known hypersensitivity to one of the trial drugs or its excipients 13. Other contraindicated concomitant treatment 14. Any condition (including drug/alcohol abuse), or laboratory results which in the investigators opinion, interfere with assessments or completion of the trial 15. Any other reason why, in the opinion of the investigator, the patient should not be enrolled in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
• Comparison of rates of sustained virologic response(SVR24) between treatment arms; defined as HCV RNA not detectable at 24 weeks after planned completion of therapy | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Nelson, Dr, Principal Investigator — St Stephens AIDS Trust, St Stephens Centre, Chelsea and Westminster Hospital, 369 Fulham Road, London, SW10 9EL
Locations (1):
- St Stephens AIDS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided